CLINICAL TRIAL: NCT01550705
Title: Quantification of the Effects of Isoniazid Treatment on Erythrocyte and Plasma Protoporphyrin IX Concentration and Plasma Aminolevulinic Acid in Patients With Erythropoietic Protoporphyria
Brief Title: Effect of Isoniazid on Protoporphyrin Levels in Erythropoietic Protoporphyria
Acronym: INHEPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis demonstrated the treatment was not effective
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Icahn School of Medicine at Mount Sinai (Other); University of Alabama at Birmingham (Other); University of California, San Francisco (Other); University of Texas (Other)
Responsible Party: Principal Investigator, John Phillips, Principle Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTINH; U54DK083909 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Erythropoietic Protoporphyria (EPP); X Linked Erythropoietic Protoporphyria
Keywords: Protoporphyria; Porphyria; Porphyrins
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Porphyrias | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Isoniazid (Experimental): Subjects will receive isoniazid daily for 2 months. Subjects will be seen every 2 weeks to obtain lab samples and health check.
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — Isoniazid 5 mg/Kg up to 300 mg per day. Oral tablets. 2 months.

SUMMARY:
In erythropoietic protoporphyria there is an accumulation of protoporphyrin IX (PPIX) in the plasma and liver. The reason it builds up is either the last step to make heme, insertion of iron into PPIX, is rate limiting or there is an increase in activity in the first step in the heme pathway.

It may be possible to decrease the amount of PPIX made and see a decrease in symptoms. The first step to make heme is the key step in the pathway and it uses vitamin B6 as a cofactor. If the investigators can limit the amount of vitamin B6 the investigators can possibly reduce the activity of this rate limiting step. With decreased activity of the enzyme it may be possible for the body to utilize all the PPIX that is made so that none builds up.

DETAILED DESCRIPTION:
Clinically, both erythropoietic protoporphyria (EPP) and X-linked EPP (XLEPP) are characterized by painful, non-blistering cutaneous photosensitivity with onset in early childhood. EPP is the most common porphyria in children and the third most common in adults (after porphyria cutanea tarda and acute intermittent porphyria). Reports of prevalence vary between 5 and 15 cases per million population.

EPP is due in most cases to decreased activity of ferrochelatase (FECH), the enzyme that catalyzes the incorporation of ferrous iron into PPIX, the final step in the production of heme. The pattern of inheritance is autosomal recessive. However, homozygosity for a FECH mutation is rare. Rather, the decreased activity is a consequence of a combination of an inherited inactivating mutation affecting one FECH allele and an intronic polymorphism that alters splicing of the other allele. The alternative splice site, when used, produces a non-functional FECH messenger ribonucleic acid (mRNA). The alternative splice site is used approximately 40% of the time. Therefore, the polymorphic allele produces approximately 60% of normal FECH activity, and for this reason, is termed hypomorphic. When the hypomorphic FECH allele is in trans with the non-functional mutant allele the result is 30% or less of the normal FECH enzyme activity. This subnormal FECH activity becomes rate-limiting, resulting in accumulation of intracellular PPIX. Although the defect is presumably expressed in all tissues, the PPIX responsible for photosensitivity derives primarily from marrow reticulocytes.

Aminolevulinic acid synthase (ALAS), the first, and rate-limiting enzyme in the heme biosynthetic pathway, catalyzes the condensation of glycine and succinyl-Coenzyme A (succinyl-CoA) to form aminolevulinic acid (ALA), and requires pyridoxal 5'-phosphate as a cofactor. ALAS in mammalian cells is localized to the mitochondrial matrix. The enzyme is synthesized as a precursor protein in the cytosol and transported into mitochondria. Two separate ALA synthase genes encode housekeeping (tissue-nonspecific) and erythroid specific forms of the enzyme (ALAS1 and ALAS2, respectively). The gene for human ALAS1 is on 3p.21 and the locus for ALAS2 the X-chromosome, at Xp11.2.

The two forms of ALAS are differentially regulated, ALAS1 is a housekeeping gene expressed in all cells and ALAS2 is driven by erythroid specific transcription factors GATA1 and NF-E2. Additionally, ALAS2 mRNA contains an iron-responsive element (IRE) in its 5'-untranslated region, similar to mRNAs encoding ferritin and the transferrin receptor (in which the IRE is in the gene's 3' UTR). Gel retardation analysis showed that the iron-responsive element in ALAS2 mRNA is functional [as evidenced by binding to iron regulator protein 2 (IRP2)], indicating that translation of the erythroid-specific mRNA is directly linked to the availability of iron and heme in erythroid cells. In this case, when intracellular iron concentration is relatively high, it is available for binding to IRP2, a process that enhances ubiquitin-mediated degradation of IRP2. Under these conditions, IRP2 is unavailable for binding to the IRE element in ALAS2, clearing the message for efficient translation. Conversely, when intracellular iron is relatively low, IRP2 degradation is restricted, making the protein available for binding to the IRE and thereby blocking translation of ALAS2 mRNA.

Recently, a variant form of EPP, inherited in an X-linked pattern (XLEPP), was shown to be due to an ALAS2 gain-of-function mutation in exon 11. The mutation results in a truncated form of the protein that has supranormal specific activity as a result of less constrained enzyme-substrate interactions, resulting in overproduction of PPIX. This situation is in contrast to EPP with mutated FECH in which PPIX accumulates because of deficient heme formation.

ALAS1 and 2 use pyridoxal phosphate (PLP) as a cofactor. PLP is a modified form of vitamin B6. It has been shown that PLP complexes with isoniazid depleting the cofactor. This PLP depletion has been one of the causes of sideroblastic anemia.

The investigators will test the hypothesis that depletion of PLP will lead to decreased activity of ALAS.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be enrolled in the Longitudinal Study of the Porphyrias.
* In patients with EPP the inclusion criteria are based on

  1. clinical features
  2. biochemical findings, as documented by laboratory reports of porphyria-specific testing performed after 1980
  3. molecular findings documenting the identification of a mutation in FECH or ALAS2 genes (molecular evidence of EPP is required for inclusion in the study).

These data will be obtained from the Porphyria Rare Disease Clinical Research Consortium Longitudinal Study (RDCRN Protocol 7201). An individual must be willing to give written informed consent and be 18 years of age or greater.

Autosomal EPP (EPP) and X-linked protoporphyria (XLEPP)

Clinical features - a or b required

* A history of non-blistering cutaneous photosensitivity, usually with early age of onset.
* A diagnosis of EPP or XLEPP in a relative.

Biochemical findings

* A marked increase in erythrocyte protoporphyrin [total erythrocyte protoporphyrin >200 ug/dL, or more than 1.5-fold increase relative to upper limit of normal of 80 ug/dL, with a predominance of free protoporphyrin (85-100% in EPP and 50-85% in XLEPP). Note: Methods in some laboratories for measuring free erythrocyte protoporphyrin (FEP) actually measure zinc protoporphyrin, so these results cannot be relied upon for diagnosis or characterizing the phenotype in EPP and XLEPP.
* Increased plasma porphyrins with a fluorescence emission peak at ~634 nm.
* Normal urinary porphyrins (except in patients with hepatobiliary impairment), and normal ALA and porphobilinogen (PBG).

Molecular findings - one of the following:

* A disease causing FECH mutation trans to the IVS3-48C>T low expression FECH allele (aEPP)
* Two disease-causing FECH mutations (EPP, recessive variant)
* A gain-of-function ALAS2 C-terminal deletion/exon 11 mutation (XLEPP)

Exclusion Criteria:

* Patients with a diagnosis of EPP that cannot be documented by DNA testing.
* Patients with evidence of active liver injury as defined by serum transaminase concentrations greater than three times the upper limit of normal, those with a history of recent (within 3 months of enrollment) or ongoing alcohol abuse, those with diabetes mellitus requiring therapy, renal insufficiency (serum creatinine >2.0 mg/ml) or evidence of malnutrition (based on subnormal plasma concentration of transthyretin) will be ineligible for participation in the study.
* Pregnant and/or lactating women will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Phillips, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: American Porphyria Foundation — http://www.porphyriafoundation.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isoniazid
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Isoniazid
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Protoporphyria Type [Count of Participants; unit: Participants]
  Erythropoietic Protoporphyria (EPP) | 9
  X-linked Erythropoietic Protoporphyria (XLEPP) | 2
Baseline Protoporphyrin IX level [Mean (Standard Deviation); unit: micrograms per deciliter (µg/dL)] | 13.3 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Protoporphyrin IX Level
Description: Plasma Protoporphyrin IX will be measured at baseline and at 3 months
Time Frame: Baseline and 3 Months
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Isoniazid
Number analyzed (Participants) | 10
µg/dL | 0.36 (9.1)

2. Secondary Outcome: Participants With Increased Sun Sensitivity
Description: Study participants were asked to report after 3 months if they had experienced an increase in subjective measures of sun sensitivity during the trial. Reported outcome is the number of study participants who reported increased sun sensitivity
Time Frame: Baseline and 3 Months
Measure: Number; unit: participants
Arm/Group | Isoniazid
Number analyzed (Participants) | 10
participants | 0

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Isoniazid
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isoniazid (N=11)
Flu-like Symptoms (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isoniazid (N=11)
Constipation (Gastrointestinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No